CLINICAL TRIAL: NCT03753815
Title: A Randomized Trial Comparing a 19-gauge EUS Fine-needle Aspiration Device With a 20-gauge Fine-needle Biopsy Device for the Diagnosis of Autoimmune Pancreatitis
Brief Title: Diagnostic Yield of FNA Needle and FNB Needle for Autoimmune Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ZS-1767
Record Dates: First submitted 2018-11-22; First posted 2018-11-27 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Autoimmune Pancreatitis
MeSH Terms: conditions — Autoimmune Pancreatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 19G FNA needle (Active Comparator): Patients referred for EUS-guided tissue acquisition of AIP
  Interventions: Device: 19G FNA needle
- 20G FNB needle (Active Comparator): Patients referred for EUS-guided tissue acquisition of AIP
  Interventions: Device: 20G FNB needle

INTERVENTIONS:
Device: 19G FNA needle — Puncture of AIP under Endoscopic Ultrasonography, with a 19-gauge FNA needle
  Other Names: 19G Echotip Ultra Fine Needle Aspiration (FNA) device
  Arms: 19G FNA needle
Device: 20G FNB needle — Puncture of AIP under Endoscopic Ultrasonography, with a 20-gauge FNB needle
  Other Names: 20G Echotip ProCore Fine Needle Biopsy (FNB) device
  Arms: 20G FNB needle

SUMMARY:
The aim of this study is to compare the diagnostic accuracy of two EUS-guided tissue acquisition devices; the 19G Echotip Ultra Fine Needle Aspiration (FNA) device and the 20G Echotip ProCore Fine Needle Biopsy (FNB) device for the diagnosis of autoimmune pancreatitis.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS)-guided tissue acquisition has emerged as a valuable method to diagnose autoimmune pancreatitis (AIP) and exclude malignancy. During Endoscopic Ultrasound (EUS), tissue samples can be obtained for pathological evaluation with different devices. Previous studies suggest 19-gauge fine needle aspiration (FNA) needle provides a reliable specimen for diagnosis of AIP. However tissue architecture and cell morphology are essential for accurate pathological assessment. Therefore, pathologists generally prefer a histological specimen. Fine needle biopsy (FNB) has the advantage of obtaining a histological specimen, which may lead to better diagnostic performance. However, the superiority of histology over cytology in EUS-guided tissue sampling for diagnosis of AIP has not been proven yet. In this study, we aim to compare the diagnostic accuracy of two EUS-guided tissue acquisition devices; the 19G Echotip Ultra Fine Needle Aspiration (FNA) device and the 20G Echotip ProCore Fine Needle Biopsy (FNB) device for the diagnosis of autoimmune pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for EUS-guided tissue acquisition because of clinical suspicion of AIP
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Known bleeding disorder that cannot be sufficiently corrected with co-fact or fresh frozen plasma (FFP)
* Use of anticoagulants that cannot be discontinued in order to guarantee an INR below 1.5
* Previous inclusion in the current study
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy (compared to the gold standard diagnosis) | 24 months
  Gold standard diagnosis is defined as: based on the conclusions of the diagnostic work-up (combined outcomes of tissue sampling and imaging studies), and confirmed by a compatible clinical disease course of at least 12 months

SECONDARY OUTCOMES:
Technical success | 24 months
  tissue acquisition
Quality of the tissue sample | within 2 weeks after the EUS procedure and after 24 months
  Quality, defined as; presence of core tissue
Quantity of the tissue sample | within 2 weeks after the EUS procedure and after 24 months
  Quantity, defined as; presence of remnant material after diagnosis was obtained and sufficiency for advanced diagnostic processing
Diagnostic yield of the first needle pass | within 2 weeks after the EUS procedure and after 24 months
Adverse events | first 24 hours until - 24 months after procedure
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Aiming Yang, M.D., Principal Investigator — Peking Union Medical College Hospitalollege Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China